CLINICAL TRIAL: NCT06502392
Title: Correlation Between Creatine Phosphokinase and Pelvic Floor Muscle Strength in Postnatal Women
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer mostafa, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/004954
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pelvic Floor; Rupture, Old (Postpartum)
Keywords: Pelvic floor strength; Creatine phosphokinase; Postnatal women
MeSH Terms: conditions — Rupture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of creatine phosphokinase — Assessment will be done through collecting a blood sample.
Other: Assessment of pelvic floor muscle strength — Assessment will be done by a biofeedback.

SUMMARY:
The purpose of this study is to determine the correlation between creatine phosphokinase and pelvic floor muscle strength in post-partum women.

DETAILED DESCRIPTION:
Pelvic floor disorders (PFDs) are complex conditions affecting women's quality of life, including issues like pelvic organ prolapse, urinary incontinence, and pelvic pain. These disorders are prevalent, with 2.6-28.7% of women experiencing urinary incontinence and 20-50% suffering from pelvic organ prolapse. Accurate diagnosis requires a comprehensive understanding of pelvic musculoskeletal components and the interaction of multiple body systems.

Creatine phosphokinase (CPK) activity can be elevated in various conditions, including muscle diseases, burns, and after strenuous exercise. During childbirth, increased serum CPK levels have been observed, attributed to enzyme release from the uterus and placenta. CPK levels typically return to normal within six weeks postpartum.

To date, no study has explored the correlation between CPK levels and pelvic floor muscle strength in postnatal women. This research aims to fill this knowledge gap, potentially benefiting medical services and expanding understanding in women's health physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Post-partum women who delivered vaginally.
* Their ages will range from 25 to 35 years old.
* Their body mass index (BMI) will be <30 Kg/m2.
* CPK will be measured within the first six weeks (2nd-5th weeks) after delivery for all women.

Exclusion Criteria:

* Any dysfunction or associated injury or any pathological conditions which may affect the result of the study as cardiac abnormalities, thyroid dysfunction recurrent urinary tract infections, uncontrolled hypertension or diabetes mellitus.
* History of pelvic inflammatory disease, myoma and tumors, pelvic infection, ovarian cyst, any gynecological disease, any hormonal abnormality and any psychological problem.
* Pelvic floor dysfunction: genital prolapse, incontinence.
* Previous surgical operations as hysterectomy.
* Inability to understand the written and verbal instructions.

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: They will be selected from the outpatient clinic of obstetrics and gynecology, Mataria Teaching Hospital, Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of creatine phosphokinase | It will be measured within the first six weeks after delivery (2nd-5th weeks).
  It will be assessed through collecting a blood sample. The collected blood will be transferred into a sterile vacutainer tubes (9 mL) with anticoagulant and will be placed symmetrically into the centrifuge device. The serum will be separated from blood and will be put in epindoorf tubes and send immediately for analysis. Serum CPK will be quantitatively measured in units/liter (u/l) on a Vitros 950 automated analyzer shortly after the receipt of the specimen.
Assessment of pelvic floor muscle strength | It will be measured within the first six weeks after delivery (2nd-5th weeks).
  It will be assessed by a biofeedback. Women will be positioned comfortably for pelvic floor muscle (PFM) strength assessment using a TG Myo feedback 420v vaginal electrode. The electrode, properly prepared and inserted, will measure vaginal closure pressure and deep PFM strength. The therapist will explain the display and will establish a one-minute baseline, noting any inconsistencies. Women will perform three 10-second maximum contractions, with the mean of these readings to be recorded. Muscle strength will be measured by peak maximum pressure and ability to sustain contraction.
Assessment of pelvic floor muscle endurance | It will be measured within the first six weeks after delivery (2nd-5th weeks).
  It will be assessed by a biofeedback. Women will be positioned comfortably for pelvic floor muscle endurance assessment using a TG Myo feedback 420v vaginal electrode. The electrode will be properly prepared and inserted. The therapist will explain the display and will establish a one-minute baseline, noting any inconsistencies. Women will perform three 10-second maximum contractions. Muscle endurance will be measured as the time a sub-maximum contraction can be maintained before significant power reduction occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Hanafy, PhD, Study Chair — Cairo University
Locations (1):
- Hadeer Mostafa, Giza, Egypt